CLINICAL TRIAL: NCT01717534
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Effect of Heat-treated Lactobacilli on Infections and Immune Status in Healthy Children
Brief Title: Children Immune Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10.42.NRC
Record Dates: First submitted 2012-10-24; First posted 2012-10-30 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Diarrhea; Upper Respiratory Infections
Keywords: Diarrhea; Children; Heat-treated lactobacilli
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heat-treated lactobacilli (Experimental): One sachets (1 gram of content) will be consumed once a day, and will be suspended in a provided milk powder to be reconstituted with water.
  The duration of the treatment is 5 months.
  Interventions: Dietary Supplement: heat-treated lactobacilli or placebo
- Maltodextrin (Placebo Comparator): One sachets (1 gram of content) will be consumed once a day, and will be suspended in a provided milk powder to be reconstituted with water.
  The duration of the treatment is 5 months.
  Interventions: Dietary Supplement: heat-treated lactobacilli or placebo

INTERVENTIONS:
Dietary Supplement: heat-treated lactobacilli or placebo — Daily supplement of sachet with 1 g of powder over a 5 months period.

SUMMARY:
The purpose of the planned study is to investigate the effect of heat-treated lactobacilli on diarrhea outcome in healthy children 1-4 years old in a randomized, double-blind, placebo-controlled study.

DETAILED DESCRIPTION:
The beneficial effect of heat-treated lactobacilli for treatment of symptomatic diarrhea was clearly documented and the purpose of this planned study is to investigate the effect on reduction of days with diarrhea in a preventive setting in healthy children 1-4 years old. Moreover, the study is intended to evaluate the impact on the immune status of the children.

ELIGIBILITY:
Inclusion Criteria:

1. Parents written and signed informed consent for participation in the study: parents agree with the participation in the study, dated and signed informed consent form prior to any study related procedure.
2. Healthy children aged 1 to 4 years
3. No more breastfed.
4. Daily home cared and going to a selected pediatrician.
5. Parents must have a phone at home or a cellular phone to call the paediatrician.
6. No consumption of commercial products containing probiotics and / or prebiotics during the 3 weeks before and during the study period.
7. Children not being intensive consumers of regular yoghurts
8. Parents are able to keep a daily record of symptoms and to administrate the study products.

Exclusion Criteria:

1. Vaccine administration within the last 3 months prior study start.
2. Used antibiotics within the last month
3. Congenital or chronic disease.
4. Any kind of immunodeficiency or allergy.
5. Acute infection or fever.
6. Significant illness within the two weeks prior to the start of the study.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 374 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Days with diarrhea | during 5 months of study period

SECONDARY OUTCOMES:
Number of episodes of upper respiratory infections | during 5 months
Duration of upper respiratory infections | during 5 months
Severity of upper respiratory infections | during 5 months
Severity of gastrointestinal infections | during 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Angeles Nava Hernández, MD, Principal Investigator — Center of Clinical Research of Querétaro; Carlos A. Mena Cedillos, MD, Principal Investigator — Clinical Research Institute
Locations (2):
- Mexico (2):
  - Clinical Research Institute, Tlalnepantla, Edo. de Méx
  - Centro de Estudios Clinicos de Queretaro S.c., Querétaro City, Querétaro